CLINICAL TRIAL: NCT01948245
Title: A Double Blinded, Randomized, Controlled Investigation of Taurolidine-citrate/Heparin Catheter Lock Solution Versus Heparin in Patients on Home Parenteral Nutrition With Previously Proven High Risk of Catheter Related Blood Stream Infections.
Brief Title: Clinical Trial Comparing Catheter Lock Solutions TaurolockTMHep 100 and Heparin 100 IE/ml.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Palle Bekker Jeppesen (Other)
Collaborators: TauroPharm (Industry)
Responsible Party: Sponsor-Investigator, Palle Bekker Jeppesen, assistent professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-4-2013-127; 38202 (Other: The National Committee on Health Research Ethics, Denmark)
Record Dates: First submitted 2013-09-16; First posted 2013-09-23 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Catheter-related Bloodstream Infection (CRBSI) Nos
Keywords: Catheter Related Blood Stream Infection; Long-term intestinal Failure; Taurolidine; Catheter lock solution; Antimicrobial agent; Home Parenteral Nutrition; Anti-infective agents
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TaurolockTMHep100 (Active Comparator): 2-4 ml of TaurolockTMHep100 will be instilled into the central venous access device (CVAD)after each infusion of parenteral nutrition/intravenous fluids. The instillation varying between twice per week to once daily depending on the patients individual HPN programme. The catheter lock solution is kept in situ in the lumen to the next infusion.
  The duration of TaurolockTMHep100 administration will be maximum 24 month or until occurence of primary outcome(CRBSI).
  Interventions: Device: TaurolockTMHep100
- Heparin 100 IE/ml (Placebo Comparator): 2-4 ml of Heparin 100 IE/mk will be instilled into the central venous access device (CVAD)after each infusion of parenteral nutrition/intravenous fluids. The instillation varying between twice per week to once daily depending on the patients individual HPN programme. The catheter lock solution is kept in situ in the lumen to the next infusion.
  The duration of Heparin 100 IE/ml administration will be maximum 24 month or until occurence of primary outcome(CRBSI).
  Interventions: Device: Heparin 100 IE/ml

INTERVENTIONS:
Device: TaurolockTMHep100 — 2-4 ml of the catheter lock solution will be instilled after each infusion of parenteral nutrition/intravenous fluids varying between twice weekly to once daily, depending on the individual patients HPN programme. The instilled solution is kept in the catheter until the next infusion, with a prior flushing with 10 ml of Saline both before the instillation of the catheter lock and before infusion of HPN/fluids.
  Other Names: Taurolidine 1,35%/citrate 4 %/heparin 100 IE/ml
  Arms: TaurolockTMHep100
Device: Heparin 100 IE/ml — 2-4 ml of the catheter lock solution will be instilled after each infusion of parenteral nutrition/intravenous fluids varying between twice weekly to once daily, depending on the individual patients HPN programme. The instilled solution is kept in the catheter until the next infusion, with a prior flushing with 10 ml of Saline both before the instillation of the catheter lock and before infusion of HPN/fluids.
  Arms: Heparin 100 IE/ml

SUMMARY:
The purpose of the investigation is to compare two catheter lock solutions (TaurolockTMHep100 and Heparin 100 IE/ml), on the occurence of catheter related blood stream infection, in patients with intestinal failure and a central venous access device for home parenteral nutrition.

DETAILED DESCRIPTION:
Patients with long-term intestinal failure are dependent on Home Parenteral Nutrition(HPN) delivered through a central venous access device(CVAD), placed as a subcutaneous tunneled catheter(Broviac). Catheter Related Blood Stream Infections(CRBSI) is a frequent complication leading to increased morbidity, hospital admissions, cost, and risk of repeated replacement of their tunneled catheter. The infections often originate from contamination of the catheter hub, and growth of microorganisms on the inner lumen of the catheter imbedded in a biofilm. To prevent infections good hygiene guidelines and the use of a catheter lock solution is applied.

The primary objective is to compare two catheter lock solutions, TaurolockTMHep100 and Heparin 100 IE/ml, on the occurence of CRBSI. The secondary objectives are to compare the two devices according to other efficacy parameters, time to infection, cost and resource utility, tolerability and safety.

Patients with a prior high risk of CRBSI will be included. Patients will instill the solution in their CVAD after each infusion of HPN, varying between minimum twice per week to once daily, depending on their individual HPN programme.

Before the blinded randomization the patients will be paired according to gender, age and prior infection risk.

Duration of the instillation will be 24 month or until outcome(CRBSI) accure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long-term intestinal failure who will receive PS at least 2 times /week over a subcutaneously tunneled single-lumen CVC (Hickman/Broviac) for at least one year.
* Estimated life expectancy ≥1 year
* Male or female patient aged 18 - 80 years
* Patient is fully able to understand the nature of the proposed intervention and gives written informed consent before entering the trial.

Exclusion Criteria:

Patients who:

* can not be expected to comply with the trial plan (e.g. substance abuse, mental condition)
* has significant cardiovascular disease such as unstable angina, recent acute myocardial infarction or recent cerebral vascular accident (within 6 weeks); a cardiac rhythm which in the investigators judgment may result in significant hemodynamic effects
* has a known hypersensitivity/allergy to TauroLockTMHep 100 or heparin and/or their excipients.
* is pregnant, lactating, or nursing
* has abnormal blood coagulation due to primary disease or due to treatment with anticoagulants (warfarin/phenprocoumon, unfractionated heparin, low- molecular heparin), with the clinical blood tests INR and APTT, outside the intervals given below, at the time of inclusion. Patients with unfractionated Heparin 100 IE/ml used as a catheter lock, do not need to have APTT tested before enrollment. Patients treated with Low-Molecular Heparin, needs control of INR, thrombocytes and plasma-antifactor Xa, and If the patient has increased bleeding risk judge by disease and clinical blood tests, the patient can´t be included in the trial. INR 0.9-3.0 (warfarin/ phenprocoumon) APTT needs to be in the range 25-100 seconds (Unfractionated Heparin treatment) Plasma-antifactor Xa( outside recommended intervals (pro.medicin.dk), which are dependent on administration form and number of daily administrations ). Thrombocytes 100- 600 x109/L
* Patients with a new catheter-related thrombosis in the last 3 months prior to inclusion.
* has received an investigational drug within 30 days of trial entry
* has received a TauroLockTMHep 100 solution previously
* has an antibiotic coated, silver impregnated or antimicrobial cuff catheter
* has compromised skin integrity, including any infection at the insertion site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mean number of catheter related blood stream infections(CRBSI)/ 1000 catheter days in each group | 24 months

SECONDARY OUTCOMES:
Median time to a catheter related blood stream infection(CRBSI) in each group. | 24 months
Number and frequency of catheter removals due to catheter-related infections in each group | 24 months
Number and frequency of exit site infections in each group | 24 months
Median time to catheter removal due to catheter-related infections in each group | 24 months
Number and frequency of catheter occlusions in each group | 24 months
Number and frequency of patients having serious adverse event and adverse event in each group | 24 months

OTHER OUTCOMES:
Patient satisfaction with the assigned catheter lock solution in each group | 24 months
  1= not at all satisfied, 2= unsatisfied, 3= satisfied, 4= very satisfied
Costs of catheter lock solution plus cost of hospitalization, unscheduled outpatient-clinic consultations, drug treatment costs of infections and catheter changes | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Palle B Jeppesen, Ass. Prof., Principal Investigator — Medicinsk Gastroenterologisk klinik CA, 2121, Abdominal centret, Rigshospitalet
Locations (1):
- Rigshospitalet, abdominalcentret, Medicinsk Gastroenterologisk klinik CA, 2121, Copenhagen, Denmark

REFERENCES:
- [Derived] Tribler S, Brandt CF, Fuglsang KA, Staun M, Broebech P, Moser CE, Scheike T, Jeppesen PB. Catheter-related bloodstream infections in patients with intestinal failure receiving home parenteral support: risks related to a catheter-salvage strategy. Am J Clin Nutr. 2018 May 1;107(5):743-753. doi: 10.1093/ajcn/nqy010. PMID 29722835
- [Derived] Tribler S, Brandt CF, Petersen AH, Petersen JH, Fuglsang KA, Staun M, Broebech P, Moser CE, Jeppesen PB. Taurolidine-citrate-heparin lock reduces catheter-related bloodstream infections in intestinal failure patients dependent on home parenteral support: a randomized, placebo-controlled trial. Am J Clin Nutr. 2017 Sep;106(3):839-848. doi: 10.3945/ajcn.117.158964. Epub 2017 Aug 9. PMID 28793993